CLINICAL TRIAL: NCT05588830
Title: The Efficacy and Safety of Telitacicept and Belimumab in Active Lupus Nephritis in the Real World: a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-353-01
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Lupus Nephritis; Belimumab; Telitacicept
MeSH Terms: conditions — Lupus Nephritis | interventions — belimumab; telitacicept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Belimumab group
  Interventions: Drug: Belimumab
- Telitacicept group
  Interventions: Drug: Telitacicept

INTERVENTIONS:
Drug: Belimumab — Belimumab, 10mg/kg, was administered intravenously on the 0, 14 and 28 days, and then once every 28 days until the 24th week
  Groups: Belimumab group
Drug: Telitacicept — Telitacicept is injected subcutaneously, 160mg/time, once a week, for a total of 24 weeks
  Groups: Telitacicept group

SUMMARY:
Lupus nephritis is an autoimmune disease. It is an inflammatory kidney damage caused by the deposition of immune complexes in the kidney. It is mainly characterized by the clinical manifestations of albuminuria, hematuria, tubular urine, pyuria, and creatinine elevation. At present, many drugs such as glucocorticoid, immunosuppressant and belimumab are used for clinical treatment, and patients still face difficulties such as complete remission, repeated relapse and so on.

This study is a multicenter, prospective, cohort study. In the study, 60 patients with lupus nephritis were enrolled, and they were treated with Telitacicept (n=30) or belimumab (n=30) for 24 weeks on the basis of conventional treatment. To observe the effectiveness and safety of the two treatment schemes for patients.

Study drug administration method:

Telitacicept was injected subcutaneously, 160mg/time, once a week, for 24 weeks.

Belimumab, 10mg/kg, was administered intravenously on the 0, 14 and 28 days, and then once every 28 days until the 24th week During the administration period of this study, the clinician fully evaluated the safety tolerance of patients using this product and decided whether to reduce the dose. The reason for adjusting the treatment plan needs to be recorded.

Reference of routine treatment plan:

High dose hormone plus cyclophosphamide was used for induction therapy, and then azathioprine or mycophenolate mofetil was used for maintenance therapy; Or high-dose hormone plus mycophenolate mofetil is used for induction therapy, and then mycophenolate mofetil is used for maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 65 years old, gender is not limited; 2. SLE patients with a clear diagnosis, that is, in line with the SLE classification criteria revised by the American College of Rheumatology in 1997 or the SLE diagnostic classification criteria issued by EULAR/ACR in 2019; 3. Patients with type III and type IV (with or without type V) lupus nephritis or simple type V lupus nephritis confirmed by biopsy within 6 months of the 2003 ISN/RPS criteria; only those with biopsy specimens showing activity were recruited Patients with lesions or active and chronic lesions; 4. ANA titer ≥ 1:80 and/or anti-dsDNA antibody positive; 5. Urine protein-to-creatinine ratio (UPCR) ≥ 1.0 mg/mg (and/or equivalent 24h urine protein level); 6. The urine protein decreased by less than 25% after receiving conventional treatment for at least 3 months before enrollment; 7. Voluntarily participate in this research and sign the informed consent.

Exclusion Criteria:

* 1. eGFR<30 mL/min/1.73m2; 2. Patients requiring dialysis or kidney transplantation; 3. Patients who have received biological agents in the past; 4. Patients who have received mesenchymal stem cell therapy in the past; 5. Those who are known to be allergic to the study drug; 6. Women who are pregnant or planning to become pregnant in the near future, and women who are breastfeeding; 7. Patients with central nervous system lupus, thrombotic microangiopathy; 8. Patients who are currently suffering from active hepatitis or have a history of severe liver disease or disease; 9. Patients with immunodeficiency, uncontrolled severe infection and active or recurrent peptic ulcer; 10. Subjects who are participating in clinical research of other drugs; In addition to the above, the investigator judges that there are other reasons for not being suitable to participate in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lupus nephritis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2023-10-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a primary renal efficacy response (PERR) | 6 months
  The main renal response response (PERR) was defined as: glomerular filtration rate (eGFR) ≥ 60ml/min/1.73m2 or eGFR decreased by no more than 20% from before recurrence; Urine protein: creatinine ratio (uPCR) ≤ 0.7; It is not a treatment failure.